CLINICAL TRIAL: NCT02533778
Title: ARISE: After 8 Hours Reperfusion in Ischemic Stroke Embolization
Acronym: ARISE
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Similar large international competing trial with results of strong positive statistically benefit
Sponsor: Abington Memorial Hospital (Other)
Responsible Party: Principal Investigator, Patricia Bussinger, MBA CRNP, Abington Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G140041
Record Dates: First submitted 2015-07-14; First posted 2015-08-27 (Estimated); Last update posted 2017-08-02 (Actual); Status verified 2017-07

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: with control group
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Interventional mechanical thrombectomy (Experimental): Mechanical thrombectomy with either Penumbra system, TREVO, or Solitaire device for acute stroke symptom onset between 8 - 24 hours
  Interventions: Device: mechanical thrombectomy

INTERVENTIONS:
Device: mechanical thrombectomy — Mechanical thrombectomy by either Penumbra system, TREVO, or Solitaire retrieval device
  Other Names: Penumbra system; TREVO; Solitaire

SUMMARY:
A prospective pilot study to evaluate the recanalization and safety of mechanical thrombectomy through a cerebral angiogram in patients with stroke symptoms last seen normal between 8 - 24 hours.

DETAILED DESCRIPTION:
Ischemic stroke patients who are 8-24 hrs from symptom onset without prior mechanical or IV thrombolytic treatment and are screen with CT or MR perfusion imaging showing penumbra and infarction not > 1/3rd the territory.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years last seen normal between 8 - 24 hours, without prior history of intravenous plasminogen activator (IV t-PA ) or
* mechanical thrombectomy Vessels - intracranial vertebral artery, basilar artery, intracranial ICA, ICA terminus bifurcation, MCA M1/M2, or
* ACA NIHSS ≥ 7 MRI DWI/PWI or
* CTA/P, which demonstrates an area of mismatch ≥ 2/3 rd
* Signed informed consent

Exclusion Criteria:

* creat >= 2
* NIHSS < 7
* Baseline mRS >= 2
* infarct > 1/3rd MCA territory
* competing trials
* prior IV or IA treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-07-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Thrombolysis in Cerebral Infarction (TICI) score | 6 months

SECONDARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) score | 6 months
Montreal Cognitive Assessment (MoCA) tool | 6 months
Modified Rankin Scale | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Qaisar Shah, MD, Principal Investigator — Abington Memorial Hospital
Locations (1):
- Abington Memorial Hospital, Abington, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided